CLINICAL TRIAL: NCT06458023
Title: Train-of-four Monitoring Using the Tetragraph Neuromuscular Transmission Monitor and Comparison to Standard (Visual) Train-of-four Assessment With a Peripheral Nerve Stimulator in Patients Less Than 1 Year of Age.
Brief Title: TOF Monitoring Using the TetraGraph in Patients Less Than 1 Year of Age
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00004121
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TetraGraph (TM) NMT Monitor (Experimental): TetraGraph is a unique, EMG-based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.
  Interventions: Device: TetraGraph (TM) NMT Monitor

INTERVENTIONS:
Device: TetraGraph (TM) NMT Monitor — TetraGraph is a unique, EMG-based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of train-of-four (TOF) monitoring using the TetraGraph Neuromuscular Transmission Monitor in pediatric patients less than 1 year of age and when feasible to compare it to standard TOF monitoring using a qualitative monitor.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-4
* ≤ 1 year of age
* undergoing a surgical procedure with general anesthesia and requiring the administration of an NMBA

Exclusion Criteria:

* Patients less than 28 days old
* Patients with history of a peripheral neurologic or neuropathic disorder
* Patients in whom the upper extremity cannot be used for TOF monitoring
* Patients undergoing a surgical procedure in which neuromuscular blockade is not required
* Edematous patients

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EMG changes | During the surgery
  Changes in the amplitude of the evoked response of the muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided